CLINICAL TRIAL: NCT03468816
Title: Clinical Functional Assessment of Moisture Sensor on Wound Dressing
Brief Title: Wound Dressing With Moisture Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vårdcentralen Åby (Other)
Collaborators: University Hospital, Linkoeping (Other); S2Clinic (Other); Absorbest AB (Other); Vinnova (Other Government); Swedish Energy Agency (Other); The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government)
Responsible Party: Principal Investigator, Fredrik Iredahl, MD, PhD., Vårdcentralen Åby
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01
Record Dates: First submitted 2018-02-26; First posted 2018-03-19 (Actual); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Ulcer, Leg; Heal Wound
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-B-A (Experimental): Investigational device is Absorbest moisture sensor in variant A and variant B, placed on the backside of the wound dressing DryMax Extra Soft. Participants performed three dressing changes. They first received variant A, at next dressing change they received variant B, and on the third dressing change they received variant A again. No washout periods.
  Interventions: Device: Sensor activation (on DryMax Extra Soft)
- B-A-B (Experimental): Investigational device is Absorbest moisture sensor in variant A and variant B, placed on the backside of the wound dressing DryMax Extra Soft. Participants performed three dressing changes. They first received variant B, at next dressing change they received variant A, and on the third dressing change they received variant B again. No washout periods.
  Interventions: Device: Sensor activation (on DryMax Extra Soft)

INTERVENTIONS:
Device: Sensor activation (on DryMax Extra Soft) — Study profile of sensor activation

SUMMARY:
Explorative study of function of a moisture sensor on top of a superabsorbent wound dressing on exuding leg ulcers.

DETAILED DESCRIPTION:
The function of a novel moisture sensor placed on a superabsorbent wound dressing has been evaluated in a small clinical investigation. Five patients with leg ulcers were included. The investigational device, Absorbest Fuktsensor, was placed on the dressing DryMax Extra Soft. Two variants of the study product were used, Variant A and Variant B. The difference between the variants were that Variant B had an extra layer of a nonwoven between the moisture sensor and the dressing in an attempt to delay the activation of the moisture sensor a little compared to Variant A which was not equipped with this nonwoven layer.

The overall aim was to observe the function of the sensor in clinical use and practical operation. Further the aim was to evaluate the two combinations of Absorbest Fuktsensor and DryMax Extra Soft and decide which combination would activate the sensor display in a satisfactory way related to the utilization of the dressings absorbing capacity while avoiding leakage and maceration.

The study was performed accordingly to ISO 14155 and the declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Presence of moderate to highly exuding leg ulcer by clinician assessment
* Wound deemed suitable for treatment with study product
* Informed consent from the participants.

Exclusion Criteria:

* Pregnancy
* Prisoner
* Bleeding from the wound
* Known allergy to components
* Wound infection
* Mental illness
* Illness or treatment of an indication other than the wound and which, according to the study personnel, can affect the wound treatment, the study and/or the dressing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD., PhD. Iredahl, Principal Investigator — Aby vardcentral, Region Ostergotland
Locations (2):
- Sweden (2):
  - Hudkliniken, University hospital, Linköping, Region Östergötland
  - S2Clinic, Linköping

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed and published on a group level.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 61 patients were screened for eligibility between May 2018 and December 2019 at the Dermatology department at University Hospital in Linköping, Sweden and 2 of these patients were enrolled.
  3 patients were screented for eligibiity and enrolled between July 2019 and December 2019 at S2Clinic in Linköping, Sweden.
Pre-assignment Details: Each enrolled participant used both investigational device Variant A and Variant B in either the order A-B-A or B-A-B according to a pre-designed schedule to ensure equal numbers in the two study arms. All 5 enrolled participants completed the study.
Period: Overall Study
Arm/Group | A-B-A | B-A-B
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A-B-A | B-A-B | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 2 | 3 | 5
Wound size [Mean (Standard Deviation); unit: cm^2] — Size of wound at inclusion of study, measured as cm2
  cm^2 | 130 (32) | 47 (17) | 80 (47)

OUTCOME MEASURES:

1. Primary Outcome: Number of Dressing Changes With Sensor Activation at Correct Timing
Description: Sensor activation - measured as indication on the sensor display; indication at correct time, indication but not att correct time, no indication.
Time Frame: Inclusion visit to study completed after 3 dressing changes, 1-2 weeks
Population: All patients recieved three dressing changes and were included in the analysis
Measure: Count of Units; unit: Dressing changes
Units Other Than Participants: Dressing changes
Groups:
- Variant A: Measure at dressing change when investigational device Absorbest moisture sensor Variant A had been used.
- Variant B: Measure at dressing change when investigational device Absorbest moisture sensor Variant B had been used.
Arm/Group | Variant A | Variant B
Number analyzed (Participants) | 5 | 5
Number analyzed (Dressing changes) | 7 | 8
Dressing changes
  Indication at correct timing | 0 | 0
  Indication, but not at correct timing | 4 | 2
  No indication | 3 | 6

2. Primary Outcome: Timing of Dressing Change Related to Dressing Size and Weight After Use
Description: Dressing weight after use were measured on a scale and recorded. The weight were compared to a predefined table.
  Dressing size 10x10 cm:
  Changed too early <11 g Correct change 11-26 g Changed too late >26 g
  Dressing size 10x20 cm:
  Changed too early <17 g Correct change 17-62 g Changed too late >62 g
  Dressing size 20x20 cm:
  Changed too early <26 g Correct change 26-109 g Changed too late >109 g
Time Frame: Inclusion visit to study completed after 3 dressing changes, 1-2 weeks
Population: All patients recieved three dressing changes and were included in the analysis.
Measure: Count of Units; unit: Dressing changes
Units Other Than Participants: Dressing changes
Arm/Group | Variant A | Variant B
Number analyzed (Participants) | 5 | 5
Number analyzed (Dressing changes) | 7 | 8
Dressing changes
  Size 10x10 cm, weight <11 g | 0 | 0
  Size 10x10 cm, weight 11 g - 26 g | 0 | 0
  Size 10x10 cm, weight >26 g | 0 | 0
  Size 10x20 cm, weight <17 g | 0 | 0
  Size 10x20 cm, weight 17 g - 62g | 3 | 6
  Size 10x20 cm, weight >72 g | 0 | 0
  Size 20x20 cm, weight <26 g | 0 | 0
  Size 20x20 cm, weight 26 g - 109 g | 3 | 0
  Size 20x20 cm, weight >109 g | 1 | 2

3. Secondary Outcome: Complications if the Dressing Was Switched Too Late.
Description: Report of leakage, strike-through and maceration at the time for dressing changes
Time Frame: Inclusion visit to study completed after 3 dressing changes, 1-2 weeks
Population: All patients recieved three dressing changes and were included in the analysis.
Measure: Count of Units; unit: Dressing changes
Units Other Than Participants: Dressing changes
Arm/Group | Variant A | Variant B
Number analyzed (Participants) | 5 | 5
Number analyzed (Dressing changes) | 7 | 8
Dressing changes
  Leakage or strike through | 3 | 2
  No leakage or strike through | 4 | 6
  Maceration due to leakage or strike through | 0 | 0

4. Secondary Outcome: Level of Usability
Description: Study the rate of handling errors
Time Frame: Inclusion visit to study completed after 3 dressing changes, 1-2 weeks
Population: All patients recieved three dressing changes and were included in the analysis.
Measure: Count of Units; unit: Dressing changes
Units Other Than Participants: Dressing changes
Arm/Group | Variant A | Variant B
Number analyzed (Participants) | 5 | 5
Number analyzed (Dressing changes) | 7 | 8
Dressing changes
  Correct application | 7 | 8
  Use errors | 0 | 0

5. Secondary Outcome: Wound Size After Three Dressing Changes
Description: Wound size after three dressing changes with the study device, measured as cm2. Can be compared with the baseline measurement of wound size.
Time Frame: At final dressing change no.3 (after 1-2 weeks)
Population: All patients recieved three dressing changes and were included in the analysis.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | A-B-A | B-A-B
Number analyzed (Participants) | 2 | 3
cm^2 | 127 (29) | 44 (16)

ADVERSE EVENTS:
Time Frame: Inclusion visit to study completed after 3 dressing changes, 1-2 weeks
Description: Adverse Event Reporting described in CIP and reported in the CRFs. All participants in the study used Variant A and Variant B at least one time.
Arm/Group | Variant A | Variant B
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Variant A (N=5) | Variant B (N=5)
Mechanical imprint (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) — Mechanical imprint from study product. Reported as mild intensity.
Adherence (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Dressing adhered to the wound. Reported as mild intensity.
Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Pain in the wound area. One report of mild pain unlikley related to the study device. One report of more pain with moderate intensity and only possibly related to the study device.
High INR value (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — High INR value in a blood sample taken between two visits. Unlikley related to the study product.
Infection (Infections and infestations) | 0 (0) | 1 (1) — Growth of Pseudomonas in wound. Graded as mild intensity and only possibly related to the study device.
Inflamed surrounding skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Inflamed surrounding skin. Graded as mild intensity and only possibly related to the study device.

LIMITATIONS AND CAVEATS:
Small trial, a first test of concept using a moisture sensor on top of a wound dressing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT03468816/Prot_000.pdf